CLINICAL TRIAL: NCT04279288
Title: The Roles of Hilotherapy in the Management of Epistaxis and Nasal Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Haroon Saeed, Specialist Trainee in ENT Surgery, Manchester University NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230638
Record Dates: First submitted 2020-02-11; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants enrolled with epistaxis and/or nasal fractures (Experimental)
  Interventions: Device: Hilotherm mask

INTERVENTIONS:
Device: Hilotherm mask — a cooling mask used to treat localized swelling and bleeding

SUMMARY:
The Investigators aimed to assess primarily whether or not Hilotherapy masks are a tolerable treatment for the conservative management of epistaxis and nasal fractures.

DETAILED DESCRIPTION:
Participants who had ongoing epistaxis and met the inclusion criteria where enrolled in the pilot study . Bleeding severity was not recorded. All participants enrolled were clinically stable with active epistaxis. Participants who were unstable or were ineligible were not referred to the recruiting doctors by A&E triage. Following informed consent the Hilotherm mask was fitted for an initial period of 20 minutes. If the bleeding had improved or stopped following 20 minutes of treatment the Hilotherm mask remained fitted for a 20 further minutes . A subjective decision was made by the supervising doctor and the participant to whether the flow of epistaxis had improved after the initial 20 minutes of hilotherapy.

The mask was removed if there was no improvement after the initial 20 minutes of hilotherapy, 40 minutes of total hilotherapy treatment, participant preference, worsening observations or profuse bleeding. Participants received conventional epistaxis management simultaneously, this involved continued nasal pressure application during hilotherapy. Following hilotherapy if epistaxis continued then either nasal cauterisation or packing was performed. Participants who were packed cessation of epistaxis was determined at the time of packing if bleeding had ceased. Bleeding time was accurately assessed by the recruiting doctor from the time of hilotherm mask application to the time of complete epistaxis cessation. All of the participants were treated in the sitting position.

Participants were free to withdraw from the trial at any time and no further data was analysed from the individual. Clinicians recorded anticoagulant and antiplatelet use, duration of bleeding and patient demographics. All participants completed a questionnaire following their hilotherapy treatment independantly.

A similar protocol was devised for nasal fractures.

ELIGIBILITY:
Inclusion Criteria:

* presenting to ED with epistaxis or nasal fractures ( over 18 years)

Exclusion Criteria:

* laceration around site of mask, reduced GCS, concurrent head injury, systemic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Outcome 1 was to assess the feasibility of using the Hilotherm mask in the first line management of epistaxis in the Accident and Emergency setting. | The outcome was measured using the patient questionnaire after the mask had been applied for 20 minutes, or in cases where epistaxis had been reduced by the mask, after 40 minutes.
  The measurement tool used to assess feasibility was a non-validated patient questionnaire. The questionnaire was provided to participants after they had worn the mask. The questionnaire was named "patient questionnaire". The questions on the questionnaire were answered by ranking choices 1 to 5. 1= strongly agree, 2= agree, 3= neither agree or disagree, 4= disagree, 5= strongly agree. The questions were as follows; The Hilotherm mask was easy to fit, The Hilotherm mask felt secure and in place, The Hilotherm mask felt comfortable to wear, the Hilotherm mask caused me discomfort/felt uncomforatble to wear, I felt the Hilotherm mask reduced the amount my nose was bleeding, I felt the Hilotherm mask was kept on for too long, if I had a nose bleed I would wear the Hilotherm mask again to reduce the bleeding.

SECONDARY OUTCOMES:
To assess the reduction in rate and severity of epistaxis when the Hilotherm mask was applied in conjunction with standard conservative measures to reduce epistaxis. | within 20 minutes of mask application
  Cessation of epistaxis was initially measured by an ENT clinician after 20 minutes of mask application. If the rate of epistaxis had reduced or the epistaxis had stopped the mask was applied for a further 20 minutes. Assessing if the epistaxis had reduced was a subjective measure, which as not based on any definable scale or units. It was depended upon the ENT doctors initial assessment of the bleeding and the resulting change in visible flow of blood from the nose after the mask had been applied. If the epistaxis has stopped this was visually defined and recorded as complete cessation of bleeding from the nose and posteriorly into the oropharynx.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No